CLINICAL TRIAL: NCT00361491
Title: An Eight-Week, Multicenter, Double-Blind, Placebo- and Paroxetine-Controlled Study Evaluating the Efficacy, and Tolerability of Two Fixed Doses of SSR149415 (250 mg Bid and 100 mg Bid) in Patients With Major Depressive Disorder
Brief Title: An Eight-Week Study Evaluating the Efficacy of Two Fixed Doses (250 mg Twice Daily and 100 mg Twice Daily) of SSR149415 in Patients With Major Depressive Disorder
Acronym: LENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI5879
Record Dates: First submitted 2006-08-07; First posted 2006-08-08 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Depressive Disorder
Keywords: Depression; antidepressive disorders; controlled clinical trial
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — 1-(5-chloro-1-((2,4-dimethoxyphenyl)sulfonyl)-3-(2-methoxyphenyl)-2-oxo-2,3-dihydro-1H-indol-3-yl)-4-hydroxy-N,N-dimethyl-2-pyrrolidinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: SSR149415

SUMMARY:
The purpose of the study is to evaluate the efficacy of SSR149415 in the treatment of Major Depressive Disorder, defined as a change from baseline to visit 7 in the Hamilton Depression Rating Scale.

To evaluate the tolerability, safety and efficacy on disability and quality of life in patients with major depressive disorder.To evaluate plasma concentrations of SSR149415.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder, recurrent, as defined by Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) criteria (296.3) and confirmed by the semi-structured Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Total score of less than 24 on the MADRS.
* HAM-D total score less than 18.
* Duration of the current depressive episode less than 1 month or greater than 2 years.
* Patients with a history or presence of bipolar disorders or psychotic disorders.
* Patients with alcohol dependence or abuse or substance dependence or abuse in the past 12 months except nicotine or caffeine dependence.
* Patients who have used the following prior to entry into Acute Phase: antipsychotics within 3 months, fluoxetine within 1 month, MAOIs within 2 weeks, other antidepressants, or mood-stabilizer (lithium, anticonvulsants) within 1 week.

The investigator will evaluate whether there are other reasons why a patient may not participate

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change from baseline to Day 56 in the 17-item Hamilton Depression Rating Scale (HAM-D) total score

SECONDARY OUTCOMES:
The main secondary endpoints are the changes from baseline to Day 56 in the HAM-D depressed mood item, Montgomery-Asberg Depression Rating Scale (MADRS) total, and Clinical Global Impression (CGI) Severity of Illness scores.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Moscow, Russia

REFERENCES:
- [Derived] Griebel G, Beeske S, Stahl SM. The vasopressin V(1b) receptor antagonist SSR149415 in the treatment of major depressive and generalized anxiety disorders: results from 4 randomized, double-blind, placebo-controlled studies. J Clin Psychiatry. 2012 Nov;73(11):1403-11. doi: 10.4088/JCP.12m07804. Epub 2012 Oct 16. PMID 23146246
- See also: Related Info — http://www.sanofi-aventis.com